CLINICAL TRIAL: NCT00689858
Title: Clinical Trial to Assessment the PK/PD Characteristics and Safety After co-Administration of Cilostazol With Ginkgo Biloba or Placebo in Healthy Subject.
Brief Title: Study to Assess the Effect of Pharmacokinetics/Pharmacodynamics (PK/PD) Interaction After co-Administration of Cilostazol With Ginkgo Biloba or Placebo
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SK Chemicals Co., Ltd. (Industry)
Responsible Party: Clinical Research Team Organization: SK Chemicals Co.,Ltd., SK Chemicals Co.,Ltd.
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GETC_DDI_I_2008
Record Dates: First submitted 2008-06-02; First posted 2008-06-04 (Estimated); Last update posted 2009-01-13 (Estimated); Status verified 2008-06

CONDITIONS: Healthy
Keywords: Healthy volunteers
MeSH Terms: interventions — Cilostazol; Ginkgo Extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): Period 1: Cilostazol, Ginkgo biloba Period 2:Cilostazol, placebo
  Interventions: Drug: Cilostazol, Ginkgo biloba and placebo
- 2 (Active Comparator): Period 1: Cilostazol, placebo Period 2: Cilostazol, Ginkgo biloba
  Interventions: Drug: Cilostazol, Ginkgo biloba and placebo

INTERVENTIONS:
Drug: Cilostazol, Ginkgo biloba and placebo — dosing time

SUMMARY:
TO assess the PK/PD effect of co-administerd Cilostazol with Ginkgo biloba or placebo, Phase I study in healthy Volunteers were designed

ELIGIBILITY:
Inclusion Criteria:

* healthy male adult volunteer between 19 and 45 years of age and within 15% of ideal body weight by broca's formula.
* the subjects who doesn't have any congenital or chronic diseases and symptoms or signs of diseases after physical examinations.]

Exclusion Criteria:

* the subject who has abnornal lab. ( In particular, AST or ALT > 1.25 times of upper limit / Total bilirubin > 1.5 times of upper limit/170,000 < Platelet < 360,000 / PT or aPTT or BT> >upper limit
* the subject who receive any metabolic enzyme inducing or inhibiting drugs like barbiturates or drink excess alcohol within 1 month prior to the study.

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2007-05; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concetration of Cilostazol at steady state | within 12hrs after cilostazol

SECONDARY OUTCOMES:
PD parameter: change from baseline after administration (change value of aggregation %) | within 12hrs after cilostazol

CONTACTS AND LOCATIONS:
Overall Officials: Jae Gook Shin, MD,PhD, Principal Investigator — Inje University
Locations (3):
- South Korea (3):
  - INJE University Pusan Paik Hospital, Pusan
  - SK chemicals, Seoul
  - SKChemicals, Seoul